CLINICAL TRIAL: NCT04883567
Title: The Use of Artificial Intelligence Real-time Feedback to Improve Compliance to a Standardised Protocol and Procedural Quality During Oesophagogastroduodenoscopy (OGD)
Brief Title: The Use of AI to Improve Quality of OGD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, CHAN SHANNON MELISSA, Assistant professor, Chinese University of Hong Kong
Other Study IDs: 2021.061
Record Dates: First submitted 2021-04-27; First posted 2021-05-12 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Dyspepsia; Anemia; Acid Reflux; Dysphagia
Keywords: oesophagogastroduodenoscopy (OGD); artificial intelligence; quality of OGD
MeSH Terms: conditions — Dyspepsia; Anemia; Gastroesophageal Reflux; Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AI arm: AI would be used to assist the trainee endoscopist
  Interventions: Diagnostic Test: The use of artificial intelligence system Cerebro
- Non-AI arm: Trainee endoscopist would perform OGD as usual.

INTERVENTIONS:
Diagnostic Test: The use of artificial intelligence system Cerebro — The artificial intelligence system Cerebro would be used during OGD
  Groups: AI arm

SUMMARY:
Early and accurate recognition of gastrointestinal lesions has implications for public health. The quality of oesophagogastroduodenoscopy (OGD) has great impact on the detection of oesophageal and gastric malignancies. An AI system, Cerebro, has been developed as a real-time recognition of a pre-defined 28 locations. This system would alert the endoscopist if the sites were not inspected with adequate time. The aim of the study is to investigate the use of AI in endoscopists-in-training during OGD to provide a real-time feedback for ensuring compliance to a standardized protocol for examination. The hypothesis is that the use of AI system Cerebro will significantly improve the compliance to the protocol and thereby reduce the blind spot rates of OGD, ensure adequate inspection time and ensure adequate photodocumentation.

ELIGIBILITY:
Inclusion Criteria:

1. All patients aged >= 18 years old
2. Undergoing diagnostic OGD for evaluation of their symptoms in the Prince of Wales Hospital will be included in the study.

Exclusion Criteria:

1. Patients in which a full endoscopic examination is not required including patients with a specific diagnostic purpose without the need for a full evaluation, follow-up endoscopy within 8 weeks for a previously diagnosed disease or condition,
2. Patients' condition requiring therapeutic endoscopy,
3. Early termination of endoscopy due to patient intolerance, presence of large amount of food residue, presence of mechanical obstruction or for reasons of safety,
4. Patients with altered anatomy such as history of esophagectomy, gastrectomy, gastric bypass surgery, or Whipple's operation,
5. Patient who are not suitable for EGD examination (such as acute peritonitis with suspected perforated bowel)
6. Pregnant females
7. Patients who refuse to participate in the study
8. Patients who are unfit for consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study includes all patients who require an OGD in the Prince of Wales Hospital. The inclusion and exclusion criteria were stated in the previous section.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
The number of sites inspected during OGD | During the procedure
  There is a standardised 28 sites the trainee endoscopist need to inspect

SECONDARY OUTCOMES:
Overall inspection time | During the procedure
  The overall inspection time during the OGD would be recorded in terms of seconds
The individual sites inspection time | During the procedure
  The individual inspection time of the 28 sites during OGD would be recorded in terms of seconds
The number of positive pathologies found on OGD | during the procedure
  The number of positive pathologies found on OGD would be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No